CLINICAL TRIAL: NCT01005472
Title: A Phase I/II Study of Daily Oral Dosing With Temozolomide and Sunitinib Malate for 6 Weeks of an 8-Week Cycle in Patients With Metastatic and Unresectable Locally-Advanced Malignant Melanoma
Brief Title: Temozolomide and Sunitinib Malate in Treating Patients With Stage III or Stage IV Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000634373; UCLA-0711052; SPRI-P05513; PFIZER-GA6181FZ; 10-001406 (Other: UCLA IRB); NCT00859326 (obsolete NCT alias)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Melanoma
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; metastatic intraocular melanoma; recurrent intraocular melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Sunitinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sunitinib malate, temozolomide (Experimental)
  Interventions: Drug: sunitinib malate; Drug: temozolomide

INTERVENTIONS:
Drug: sunitinib malate
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving temozolomide together with sunitinib malate may kill more tumor cells.

Phase II was never conducted due to toxicity in phase I.

PURPOSE: This phase I/II trial is studying the side effects and best dose of sunitinib malate when given together with temozolomide and to see how well they work in treating patients with stage III or stage IV malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the maximum tolerated dose of sunitinib malate when administered concurrently with temozolomide in patients with stage IIIC or IV malignant melanoma. (Phase I)
* Assess the overall safety of this regimen in these patients. (Phase I)
* Determine the response rate in patients treated with this regimen. (Phase II) Phase II was never conducted due to toxicity in phase I.

Secondary

* Determine the response rate in patients treated with this regimen. (Phase I)
* Determine the safety and tolerability of this regimen in these patients. (Phase II)
* Determine the progression-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a phase I, dose-escalation study of sunitinib malate followed by a phase II study.

Patients receive oral sunitinib malate once daily and oral temozolomide once daily on days 1-42. Treatment repeats every 56 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up very 6 months for up to 5 years.

Phase II was never conducted due to toxicity in phase I.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage IIIC unresectable cutaneous or mucosal melanoma with measureable disease or stage IV cutaneous, mucosal or ocular melanoma with measureable disease.
* ECOG performance status of 0-2
* age greater than or equal to 18 years
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Hemoglobin ≥ 10.0 g/dL
* Creatinine ≤ 2 times upper limit of normal (ULN)
* Total bilirubin ≤ 2 times ULN
* LDH ≤ 5 times ULN
* AST or ALT ≤ 2.5 times ULN (≤ 5 times ULN if liver metastasis is present)
* LVEF ≥ 50% on screening ECHO
* women of childbearing potential must have a negative urine or serum pregnancy test upto 28 days prior to commencement of dosing.
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* before study entry , written informed consent must be obtained. Written informed consent must be obtained from patient prior to performing any study related procedures.

Exclusion Criteria

* pregnant or nursing
* any following within the past 12 months:
* Myocardial infarction
* Severe and/or unstable angina
* Coronary and/or peripheral artery bypass graft
* Symptomatic congestive heart failure
* Cerebrovascular accident or transient ischemic attack
* Pulmonary embolism
* ongoing cardiac dysrhythmias ≥ grade 2, according to NCI CTCAE v3.0
* prolonged QTc interval on baseline EKG
* uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg despite optimal medical therapy)
* pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* any known clinically uncontrolled infectious disease, including HIV positivity or AIDS-related illness
* severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results, and, in the judgment of the investigator, would make the patient inappropriate for study entry
* prior chemotherapy for melanoma, except for chemotherapy given during isolated limb perfusion for stage IIIC disease
* Prior adjuvant immunotherapy and/or immunotherapy for metastatic disease allowed
* prior major surgery, radiotherapy, or immunotherapy within 4 weeks of starting therapy
* treatment with potent CYP3A4 inhibitors 7 days before study dosing
* treatment with potent CYP3A4 inducers 12 days before study dosing
* concurrent treatment on another clinical trial (Concurrent participation on supportive care trials or non-treatment trials (e.g., quality-of-life trials) allowed).
* concurrent chemotherapy, immunotherapy, biological therapy, or investigational drugs
* concurrent drugs with dysrhythmic potential, including any of the following:
* Terfenadine
* Quinidine
* Procainamide
* Disopyramide
* Sotalol
* Probucol
* Bepridil
* Haloperidol
* Risperidone
* Indapamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of sunitinib malate when administered concurrently with temozolomide (Phase I) | 6 weeks
Overall safety | 5 years
Response rate as assessed by modified RECIST criteria (phase II) | 5 years
  Phase II was never conducted due to toxicity in phase I.

SECONDARY OUTCOMES:
Response rate as assessed by modified RECIST criteria (Phase I) | 6 weeks
Progression-free survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Chmielowski, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles (UCLA), Los Angeles, California, United States